CLINICAL TRIAL: NCT03399123
Title: Effect of Low Tidal Volume on Blood Loss During Laparoscopic Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Institute of Hepatobiliary Surgery, Southwest Hospital, Third Military Medical University Affiliation: Southwest Hospital, China, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MZK001
Record Dates: First submitted 2018-01-04; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Blood Loss
Keywords: Laparoscopic hepatectomy; Low tidal volume; Blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tidal Volume

STUDY DESIGN:
Intervention Model Description: Two different tidal volume are conducted on the participant base on the randomized choices
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low tidal volume group (Experimental): Use a low tidal volume(6'8ml/kg) ventilation mode during liver segmentation。
  Interventions: Other: Tidal volume
- Standard tidal volume group (Active Comparator): Use a standard tidal volume(10'12ml/kg) ventilation mode during operation.
  Interventions: Other: Tidal volume

INTERVENTIONS:
Other: Tidal volume — After General anesthesia, patients that during volume control mode of mechanical ventilation in experimental group, we take low tidal volume.

SUMMARY:
To explore the effect of low tidal volume on blood loss and gas exchange during laparoscopic hepatectomy

DETAILED DESCRIPTION:
Background & Aims:Liver cancer is an disease that threatening human health .Laparoscopic hepatectomy is more and more widely used.It is very important to reduce the bleeding during laparoscopic hepatectomy.The investigators found that low tidal volume can effectively reduce intraoperative bleeding.The aim of this study was to explore the effect of low tidal volume on blood loss and gas exchange during laparoscopic hepatectomy

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 70 years old;
2. American association of anesthesiologists(ASA) score I to III;
3. Ability to adhere to the study schedule;
4. Ability to provide informed consent and complete all study assessments;
5. Patients undergoing selective surgery of laparoscopic hepatectomy.

Exclusion Criteria:

1. The New York Heart Association classification(NYHA) III to IV;
2. Chronic obstructive pulmonary disease,respiratory failure, patients after thoracic surgery.
3. BMI>32Kg/m2;
4. Abnormal in blood coagulation function;
5. Patients with mental disease;
6. Patients with neuromuscular disease;
7. Concurrent enrollment in another Randomized controlled trial(RCT);
8. Absence of written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Blood loss | through study completion, an average of 48hours
  Blood loss during operation.

SECONDARY OUTCOMES:
central venous pressure | During operation
  The central venous pressure(CVP)during operation
mean arterial pressure | During operation
  The mean arterial pressure(MAP)during operation
oxygenation index | During operation
  The oxygenation index during operation.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng ShuGuo, Principal Investigator — MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China